CLINICAL TRIAL: NCT00193284
Title: A Phase I/II Trial of Induction Chemotherapy Plus Gefitinib (Iressa) Followed by Concurrent Chemotherapy, Radiation Therapy, and Gefitinib (Iressa) For Patients With Locally Advanced Squamous Carcinoma of the Head and Neck
Brief Title: Chemotherapy Plus Gefitinib Followed by Chemotherapy, Radiation Therapy, and Gefitinib For Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: AstraZeneca (Industry); Aventis Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI HN 04; IRUSIRES0047; IIT 15038
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gefitinib; Docetaxel; Carboplatin; Fluorouracil

INTERVENTIONS:
Drug: Gefitinib
Drug: Docetaxel
Drug: Carboplatin
Drug: Fluorouracil

SUMMARY:
Although gefitinib has been combined successfully with various chemotherapeutic regimens with minimal increase in overall toxicity, experience with concurrent radiation therapy is limited. In this trial, we will evaluate the feasibility, toxicity, and effectiveness a novel combination of chemotherapy, radiation therapy, and gefitinib.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will receive:

Induction Therapy

* Docetaxel
* Carboplatin
* 5-FU
* Gefitinib

Combined Modality Therapy

Cohort 1:

* Radiation therapy
* Gefitinib

Cohort 2:

* Radiation therapy
* Gefitinib
* Docetaxel

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Squamous carcinoma of the head and neck.
* Primary tumor nasopharynx, oral cavity, oropharynx, hypopharynx, and larynx
* Squamous carcinoma in cervical nodes no identified primary site
* Must be considered to have low cure rates with local therapy
* Previously untreated with chemotherapy or radiation therapy.
* Able to perform activities of daily living without assistance
* Adequate bone marrow, liver, and kidney function
* Mild peripheral neuropathy is allowed
* Measurable or evaluable disease
* Voluntarily give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* History of prior malignancy within the last five years
* Severe or uncontrolled systemic disease
* Significant clinical disorder or laboratory finding
* Women who are pregnant or breast-feeding
* Active interstitial lung disease

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-10; Primary Completion 2006-02 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Overall survival
Time to progression
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Burris HA 3rd, Markus TM, Shipley D, Kuzur M, Lunin S, Greco FA. Neoadjuvant chemotherapy/gefitinib followed by concurrent chemotherapy/radiation therapy/gefitinib for patients with locally advanced squamous carcinoma of the head and neck. Cancer. 2009 May 15;115(10):2138-46. doi: 10.1002/cncr.24265. PMID 19288572